CLINICAL TRIAL: NCT06768684
Title: Alcohol Related Risk Reduction in Rural Veterans
Brief Title: Alcohol Related Risk Reduction in Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Vander Weg, Investigator, Iowa City Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOMAD 4130
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use
Keywords: alcohol; harm reduction; behavioral intervention; Veterans
MeSH Terms: conditions — Alcohol Drinking; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active intervention (Experimental): Veterans will receive a two-session telephone-administered alcohol risk reduction intervention.
  Interventions: Behavioral: Brief behavioral counseling

INTERVENTIONS:
Behavioral: Brief behavioral counseling — Participants receive a two-session phone-based alcohol risk reduction intervention based on principles of harm reduction. Participants receive personalized feedback regarding how alcohol use may impact their health. Following a motivational enhancement exercise, participants are advised to reduce alcohol intake to within recommended limits. Evidence-based strategies are discussed (e.g., goal setting, self-monitoring, identifying and avoiding triggers, dealing with urges, pacing and spacing drinks, managing high risk situations, finding alternatives to alcohol, developing refusal skills, and enlisting social support). Educational materials addressing methods for cutting down are also provided, along with information about other available resources to support their efforts.

SUMMARY:
This project is designed to refine and evaluate the feasibility and preliminary effectiveness of a brief, telephone-administered alcohol risk reduction intervention for Veterans.

DETAILED DESCRIPTION:
This study will investigate whether a brief alcohol harm reduction intervention for Veteran primary care patients who consume alcohol at levels that exceed dietary guidelines but who do not necessarily exhibit evidence of alcohol use and dependence is feasible based on enrollment and retention rates, and treatment satisfaction. In addition, we will investigate whether there is preliminary evidence for efficacy of the intervention based on changes in alcohol consumption over time.

Following enrollment in the study, participants will be scheduled for an initial phone session. Veterans will then receive an alcohol risk reduction intervention that is based on VA/DoD Clinical Practice Guidelines and strategies recommended by the National Institute on Alcohol Abuse and Alcoholism (NIAAA). The intervention will be delivered via telephone. After an introduction and overview of the intervention, Veterans will be provided with personalized feedback regarding potential health risks associated with their alcohol use and how alcohol use may interact with their health conditions and medications. Following a motivational enhancement exercise, Veterans are advised to reduce alcohol intake to within recommended limits and are supported in identifying a drinking goal. Consistent with principles of harm reduction, the approach starts by "meeting the Veteran where they are" and establishing a collaborative and empowering relationship that leverages the individual's skills. Rather than requiring participants to work toward abstinence, Veterans select their own treatment goals. Evidence-based strategies for achieving the goal are discussed (e.g., goal setting, self-monitoring, identifying and avoiding triggers, dealing with urges, pacing and spacing drinks, managing high risk situations, finding alternatives to alcohol, developing refusal skills, and enlisting social support). Educational materials addressing methods for cutting down are also provided, along with information about other available resources to support their efforts. Progress is monitored at a subsequent contact. Small, incremental gains are reinforced and recognized as steps in the right direction. Problem solving is used to address barriers to change, and revised goals are discussed as appropriate.

Participants will complete baseline questionnaires as well as a post-treatment evaluations (at approximately three months) and follow-up questionnaires at six months post baseline. Data collection will occur by phone unless the participant requests a hard copy survey to be mailed.

Some study participants will also be selected for a separate phone call to ask additional questions about their experience with the coaching sessions, such as what they liked and didn't like about the phone calls, and what things about them were the most and least helpful.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status, English-speaking, report current alcohol use, receiving treatment through the Iowa City VA Health Care System

Exclusion Criteria:

* History of significant alcohol withdrawal, evidence of significant alcohol dependence, lack of regular access to a telephone, inability to participate in phone counseling

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | 30-days
  Past 30-day alcohol consumption will be assessed using the Alcohol Timeline Follow-back method.

IPD SHARING:
Plan to Share IPD: Undecided